CLINICAL TRIAL: NCT06806813
Title: Italian Anderson Fabry Disease Cardiovascular Registry
Acronym: RICMAF
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: RICMAF
Record Dates: First submitted 2025-01-09; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-11

CONDITIONS: Fabry Disease
Keywords: Fabry
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The RICMAF Study is an observational, multicenter, non-pharmacological study conducted in Italy.

Although Anderson-Fabry Disease (AFD) is rare, it is likely underdiagnosed due to its nonspecific symptoms, leading to delays in proper treatment. The RICMAF Study aims to improve understanding of AFD, especially its cardiac manifestations, which are a major cause of mortality. By gathering data from a large, nationwide patient registry, this study seeks to answer key questions about AFD's clinical course and improve patient outcomes.

The primary goals of the RICMAF Study are:

* To analyze the clinical profile, prevalence, and incidence of AFD, along with patients' family history and disease progression.
* To identify early markers of cardiac involvement and predictors of cardiovascular complications to personalize care.
* To investigate the relationship between genetic mutations, clinical presentation, and prognosis.
* To find early indicators of organ damage through laboratory and imaging tests.

All patients diagnosed with AFD following international guidelines are eligible.

DETAILED DESCRIPTION:
1. Introduction

   Anderson-Fabry Disease (AFD) is a multisystemic lysosomal storage disorder with X-linked inheritance (Online Mendelian Inheritance in Man [OMIM] number 301500) caused by a total or partial deficiency of the enzyme α-galactosidase A (α-Gal A), encoded by the GLA gene (Xq22.1). The deficiency of α-Gal A leads to the accumulation of neutral glycosphingolipids, particularly globotriaosylceramide (Gb3) and galactosylceramide, in various cell types and tissues. The continuous accumulation of these molecules results in progressive cellular dysfunction, triggering inflammatory and pro-fibrotic phenomena that cause organ dysfunction.

   The clinical manifestations and age of onset of the disease are highly variable, and symptoms/signs often appear only after a degree of irreversible damage has already occurred. The classic form of AFD is the most severe clinical phenotype and predominantly affects males with null or minimal residual enzymatic activity (<1% of normal values). Symptoms begin early during childhood or adolescence and include acroparesthesias, angiokeratomas, telangiectasias, gastrointestinal disturbances, corneal alterations (cornea verticillata), proteinuria, renal insufficiency, hypo/hyperhidrosis, and hearing loss. Later in adulthood, progressive cardiac and cerebrovascular involvement may occur.

   Patients with atypical or late-onset variants generally develop the disease later (from the third to the seventh decade of life) compared to those with the classic form. The clinical picture is generally dominated by the involvement of a single organ, most frequently the heart. The measurement of residual enzymatic activity of α-Gal A is sufficient to establish a diagnosis in males. However, it is important to identify the specific genetic mutation to determine the disease phenotype and exclude benign polymorphisms that may cause reduced enzymatic activity levels. In females, genetic diagnosis is indispensable, as residual enzymatic activity often falls within the normal range.

   The treatment of AFD is based on compensating for the deficient enzymatic activity through enzyme replacement therapy (ERT) and managing the disease's symptoms and complications. More recently, an oral chaperone therapy capable of increasing residual enzymatic activity has been approved, though it is only effective for certain mutation types. Given the multisystemic involvement in AFD patients, longitudinal multispecialty evaluation is necessary, including cardiology, nephrology, neurology, dermatology, ophthalmology, and otorhinolaryngology assessments.

   Cardiac involvement is the main prognostic factor, with cardiovascular death being the leading cause of mortality. Manifestations include unexplained ventricular hypertrophy (which must be differentiated from the more common sarcomeric hypertrophic cardiomyopathy), valvular diseases, angina pectoris due to coronary microcirculation dysfunction, conduction abnormalities (which may require permanent pacemaker implantation), and supraventricular and ventricular tachyarrhythmias. Cardiological evaluation is recommended annually or earlier if clinically indicated, including systemic blood pressure assessment, ECG, echocardiography, and arrhythmia detection via 24-hour Holter ECG monitoring (or extended monitoring [e.g., loop recorder] when deemed appropriate).

   In recent years, cardiac magnetic resonance imaging (CMR) has become a key investigation not only for diagnosing the disease but also for its follow-up and for evaluating the response to therapy. CMR allows for accurate assessment of cardiac chamber volumes and function and enables tissue characterization using gadolinium-based contrast agents and advanced T1 and T2 mapping techniques. Endomyocardial biopsy is now reserved for patients with genetic variants of uncertain significance (VUS), high residual enzymatic activity (>10%), and/or low lyso-Gb3 levels to confirm or exclude AFD as the cause of left ventricular hypertrophy.
2. Study Background

   AFD is a rare disease, and the estimated prevalence of the classic forms was previously reported to range between 1:40,000 and 1:117,000. However, these data likely represent an underestimation, as the manifestations are nonspecific, and AFD is often not considered among diagnostic hypotheses, leading to misdiagnosis or delayed diagnosis. Supporting this, recent genetic newborn screening programs not based on symptom development suggest that AFD may be far more common than previously suspected.

   Although the last decade has seen increasing understanding of the disease's pathophysiological mechanisms, natural history, and the efficacy and limitations of current therapeutic options, many unanswered questions remain. This highlights the need to create an Italian cardiological registry for Anderson-Fabry Disease to bring together various centers located in different regions nationwide to collect the largest possible number of patients.
3. Study Objectives

   * Evaluate the clinical profile, prevalence, and incidence of the disease (relative to the general population), as well as the family and natural history of AFD patients, particularly the incidence of morbidity/mortality during follow-up.
   * Identify clinical and instrumental predictors of cardiovascular morbidity and mortality to improve risk stratification and personalize the most appropriate management program for each patient.
   * Assess the correlation between genetic findings, phenotype, and prognosis, with particular emphasis on differences in cardiac involvement between classic and late-onset variants with cardiac involvement.
   * Investigate serological/tissue markers and instrumental indicators of early organ damage.
4. Study Plan

   4.1 Study Population All patients affected by Anderson-Fabry Disease (AFD), diagnosed according to current international guidelines, will be included in the study upon obtaining informed consent. Based on the estimated prevalence of the disease, the study plans to enroll approximately 800 patients over 10 years.

   Inclusion Criteria:
   * Patients diagnosed with Anderson-Fabry Disease.
   * Age ≥ 2 years at the time of diagnosis.
   * Informed consent obtained from the patient or their parent/legal guardian.

   Exclusion Criteria:

   - None.

   4.2 Study Design

   The study is an Italian multicenter, observational, retrospective, and prospective, non-pharmacological study. Participation will be proposed consecutively to all patients with AFD attending the participating centers, both as outpatients and inpatients.

   Structured data collection for objective evaluation will occur through a dedicated electronic archive, gathering data from the observation period between January 1, 1981, and December 31, 2031. This electronic archive may be used to obtain or confirm new scientific evidence regarding AFD, particularly focusing on diagnosis, prognosis, and therapy.

   Data entry into the electronic archive will be based on the review of medical records (outpatient or inpatient), collecting information about demographics, past and recent medical history, family history, genetic investigations, instrumental assessments, signs and symptoms of the disease, and therapy.

   Data Collection Modes:
   * Prospective Phase: Patients will be enrolled during hospitalization or at the first outpatient visit after obtaining free and informed consent. Patients will subsequently undergo clinical evaluations, instrumental investigations, and therapeutic interventions as per clinical necessity and standard care practices. A minimum follow-up duration is not required; even a single evaluation suffices for inclusion in the archive.
   * Retrospective Phase: Data from patients will be retrospectively collected starting from January 1, 1981. In this phase, no predefined observation period is required. If the patient is no longer being followed, a substitute declaration of consent for retrospective observational studies will be used to utilize clinical/instrumental data excluding genetic data.

   In all cases where it is possible to provide adequate information, particularly when patients return to care centers for health services or follow-up visits, their consent for data processing must be obtained.

   4.3 Discontinuation of Participation

   Patients may choose to discontinue their participation in the study at any time.

   4.4 Visits and Assessments

   Specialist visits, laboratory tests, genetic analyses, and instrumental evaluations to which patients are or will be subjected fall within the normal care pathway, in line with the standard of care. The data collected will derive from initial and follow-up visits or hospitalizations that are part of standard clinical practice.
5. Data Management and Statistical Analysis

   5.1 Data Collection Methods Systematic data collection will occur through the creation of a dedicated electronic archive, collecting data for the observation period between January 1, 1981, and December 31, 2031. Clinical data required by the protocol will be pseudonymized and entered by designated staff into an electronic Case Report Form (eCRF) managed via the REDCap platform. The eCRF in REDCap will be developed and managed following the procedure outlined in the "Operational Instruction for the Management and Use of the REDCap Platform" (IOA119).

   The Principal Investigator must specify the personnel delegated for data management and their respective roles in the study in the Delegation Log. Collected data will be derived from standard care medical records, with no study-specific assessments performed.

   5.2 Statistical Methods The collected data will include demographics (age, gender), medical history, instrumental data (ECG, echocardiography, cardiac MRI, stress tests, 24-hour Holter ECG, biopsies), laboratory data (CBC, platelets, renal and liver function, BNP, troponin, serum electrolytes, urinalysis, etc.), genetic investigation findings, and follow-up data.

   The results of the analysis will be processed statistically in anonymous form to derive the study objectives. Data will be presented using descriptive statistics:
   * Qualitative parameters will be expressed as numbers or percentages and analyzed using Chi-square or Fisher's exact test.
   * Quantitative parameters will be expressed as mean and standard deviation or as median and interquartile range, with comparisons between patients performed using parametric tests (ANOVA, Student's t-test) or non-parametric tests (Kruskal-Wallis and Mann-Whitney U tests).

   A p-value ≤ 0.05 will be considered statistically significant. Statistical analyses will be conducted using Stata/SE v.14.2 for Windows.
6. Administrative Procedures

Good Clinical Practice Guidelines This study will be conducted in compliance with Good Clinical Practice (GCP) guidelines [ICH Harmonized Tripartite Guidelines for GCP 1996 Directive 91/507/EEC; D.M. 15.7.1997], the Declaration of Helsinki, and national regulations governing clinical research. By signing the protocol, the investigator agrees to adhere to the procedures and instructions contained therein and to conduct the study according to GCP, the Declaration of Helsinki, and national regulations on clinical trials.

Protocol Amendments or Study Modifications Any protocol modifications will be implemented as formal amendments. No protocol modifications are allowed during the study period. Any unforeseen changes in study conduct will be documented in the "Clinical Study Report."

Ethical Committee Approval The study protocol, any amendments, informed consent forms, and patient information must be approved by the Ethics Committee. For amendments, the Investigator may immediately implement changes to ensure patient safety and must notify the Ethics Committee within 10 working days.

Consent Management Patients will be enrolled during hospitalization or outpatient visits, and each participant must sign an informed consent form.

* For the prospective phase, consent will be obtained during the standard diagnostic process.
* For the retrospective phase, concerning previously collected data, informed consent will be sought during follow-up visits. For deceased or unreachable patients, data will be processed without consent based on General Authorization No. 146/2019 from the Privacy Authority, excluding genetic data.

Documentation Archive.

The Investigator is responsible for archiving and storing essential study documents before, during, and after the study in compliance with applicable regulations and GCP. Data in the CRF will be strictly anonymous, and subjects will be identified only by a number and initials.

Publication of Results Data publication will occur after processing during the data collection period or after the final update of the archive.

Costs No additional costs are foreseen for conducting this study. Clinical evaluations and instrumental examinations are routinely performed in these patients as part of standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Anderson Fabry disease
* Age ≥ 2 years at diagnosis
* Obtaining informed consent from the patient and parent or legal guardian.

Exclusion Criteria:

- None

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients affected by AFD, diagnosed according to current international guidelines, will be included in the study, after obtaining free and informed consent. The study plans, based on the estimated prevalence of the disease, to enroll approximately 800 patients over the course of 10 years.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-01-26 (Actual); Primary Completion 2031-01-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Definition of Fabry disease natural history | From enrollment to mean follow-up of 5 years.
  * Prevalence of Fabry disease: number of diagnosed cases of Fabry disease per 100,000 individuals in the general population.
  * Incidence of Fabry disease: number of new cases of Fabry disease per year per 100,000 individuals in the general population.
  * Number of patients with morbidity (heart failure, arrhythmias, kidney failure, stroke) and mortality (cardiac and non cardiac death) events recorded during follow-up.

SECONDARY OUTCOMES:
Fabry disease cardiac risk stratification | From enrollment to mean follow-up of 5 years.
  To identify clinical and instrumental predictors of morbidity and cardiovascular mortality, in order to enhance risk stratification of events and to personalize the most appropriate management plan for each patient.
Correlation between genotype and cardiac involvement (ECG changes, LVH, T1/T2 mapping)/cardiac events. | From enrollment to mean follow-up of 5 years.
  To assess the correlation between genetic results (missense vs non-missense variants), phenotype (ECG abnormalities, degree of LVH by echo/CMR; T1 and T2 mapping values by CMR; amount of scar [LGE] by CMR) ), and prognosis (mortality/morbidity), with particular focus on differences in cardiac involvement between classic and late-onset forms with cardiac involvement.
Identification of biomarkers for early diagnosis in Fabry disease | From enrollment to mean follow-up of 5 years.
  To investigate serological/tissue markers (troponin [ng/L], BNP [pg/L], microRNA [copies/ml]] and instrumental indicators (vacuolization by histology, T1 an T2 values by CMR) of early cardiac damage.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Biagini, MD, PhD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (54):
- Italy (54):
  - ASL 2 Chieti - Ospedale Policlinico SS. Annunziata, Chieti, Abruzzo/Chieti
  - Azienda Ospedaliera Regionale S.Carlo, Potenza, Basilicata/Potenza
  - AORN "Sant'Anna e San Sebastiano" di Caserta, Caserta, Caserta
  - Azienda Ospedaliero - Universitaria "Mater Domini, Catanzaro, Catanzaro
  - Azienda Ospedaliera di Cosenza Università della Calabria, Cosenza, Cosenza
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, EmiliaRomagna/Bologna
  - IRCCS Ospedale Policlinico San Martino, Genova, Genova
  - ASST Papa Giovanni XXIII, Bergamo, Lombardia/Bergamo
  - U.O.Cardiologia Spetali Civili 1, Brescia, Lombardia/Brescia
  - IRCCS Ospedale Maggiore Policlinico di Milano, Milan, Lombardia/Milano
  - IRCCS San Gerardo dei Tintori - S.C. Nefrologia, Monza - Università di Milano Bicocca, Milan, Lombardia/Milano
  - Centro Cardiologico Monzino, Milan, Lombardia/Milano
  - Ospedale Niguarda, Milan, Lombardia/Milano
  - IRCCS Policlinico San Donato, San Donato Milanese, Lombardia/Milano
  - A O Universitaria Ospedali Riuniti Ancona, Ancona, Marche/Ancona
  - Clinica cardiologica AZ ospedaliera Torrette, Ancona, Marche/Ancona
  - AO Dei Colli - Ospedale Monaldi, Napoli, Napoli
  - AOU Policlinico, Napoli, Napoli
  - Azienda Ospedaliero-Universitaria di Parma, Parma, Parma
  - Azienda Ospedaliera "Guglielmo da Saliceto" di Piacenza, Piacenza, Piacenza
  - Ospedale Ivrea, Ivrea, Piemonte/Ivrea
  - Ospedale Maggiore della Carità, Novara, Piemonte/Novara
  - Molinette, Torino, Piemonte/Torino
  - Ospedale Koelliker di Torino, Torino, Piemonte/Torino
  - Policlinico Bari, Bari, Puglia/Bari
  - A O Universitaria Ospedali Riuniti di Foggia, Foggia, Puglia/Foggia
  - Ospedale Casa Sollievo della sofferenza, Manfredonia, Puglia/Foggia
  - Ospedale Vito Fazzi, Lecce, Puglia/Lecce
  - Ospedale SS.ma Annunziata, Taranto, Puglia/Taranto
  - Ospedale Metropolitano Riuniti "Bianchi - Melacrino - Morelli, Reggio Calabria, Reggio Calabria
  - Arcispedale S.Maria Nuova, Reggio Emilia, Reggio Emilia
  - Ospedale degli Infermi di Rimini, AUSL Romagna, Rimini, Rimini
  - Policlinico "Tor Vergata", Roma, Roma
  - Policlinico Gemelli, Roma, Roma
  - Policlinico Umberto I - Università Sapienza, Roma, Roma
  - Policlinico Casilino, Roma, Roma
  - Ospedale Sant'Andrea, Roma, Roma
  - San Camillo Forlanini, Roma, Roma
  - Ospedale S.Giovanni di Dio e Ruggì d'Aragona, Salerno, Salerno
  - Azienda Ospedaliera G. Brotzu, Cagliari, Sardegna/Cagliari
  - Azienda Ospedaliera Universitaria, Cagliari, Sardegna/Cagliari
  - Policlinico Rodolico, Catania, Sicilia/Catania
  - Policlinico G. Martino, Messina, Sicilia/Messina
  - Policlinico P. Giaccone, Palermo, Sicilia/Palermo
  - Ospedale San Donato, Arezzo, Toscana/Arezzo
  - Azienda Ospedaliero Universitaria Careggi e Meyer, Florence, Toscana/Firenze
  - Fondazione Toscana Gabriele Monasterio, Pisa, Toscana/Pisa
  - Azienda Ospedaliera Universitaria Siena, Siena, Toscana/Siena
  - Ospedale S.Chiara, Trento, Trentino Alto Adige/Trento
  - Azienda sanitaria universitaria Giuliano Isontina, Trieste, Triesta
  - Azienda sanitaria universitaria Friuli Centrale, Udine, Udine
  - Ospedale di Perugia, Perugia, Umbria/Perugia
  - Ospedale Padova, Padua, Veneto/Padova
  - Ospedale Policlinico Sede di Borgo Roma, Verona, Veneto/Verona

REFERENCES:
- [Background] Nordin S, Kozor R, Medina-Menacho K, Abdel-Gadir A, Baig S, Sado DM, Lobascio I, Murphy E, Lachmann RH, Mehta A, Edwards NC, Ramaswami U, Steeds RP, Hughes D, Moon JC. Proposed Stages of Myocardial Phenotype Development in Fabry Disease. JACC Cardiovasc Imaging. 2019 Aug;12(8 Pt 2):1673-1683. doi: 10.1016/j.jcmg.2018.03.020. Epub 2018 May 16. PMID 29778854
- [Background] Pieroni M, Moon JC, Arbustini E, Barriales-Villa R, Camporeale A, Vujkovac AC, Elliott PM, Hagege A, Kuusisto J, Linhart A, Nordbeck P, Olivotto I, Pietila-Effati P, Namdar M. Cardiac Involvement in Fabry Disease: JACC Review Topic of the Week. J Am Coll Cardiol. 2021 Feb 23;77(7):922-936. doi: 10.1016/j.jacc.2020.12.024. PMID 33602475
- [Background] Linhart A, Germain DP, Olivotto I, Akhtar MM, Anastasakis A, Hughes D, Namdar M, Pieroni M, Hagege A, Cecchi F, Gimeno JR, Limongelli G, Elliott P. An expert consensus document on the management of cardiovascular manifestations of Fabry disease. Eur J Heart Fail. 2020 Jul;22(7):1076-1096. doi: 10.1002/ejhf.1960. Epub 2020 Aug 14. PMID 32640076
- [Background] Germain DP, Hughes DA, Nicholls K, Bichet DG, Giugliani R, Wilcox WR, Feliciani C, Shankar SP, Ezgu F, Amartino H, Bratkovic D, Feldt-Rasmussen U, Nedd K, Sharaf El Din U, Lourenco CM, Banikazemi M, Charrow J, Dasouki M, Finegold D, Giraldo P, Goker-Alpan O, Longo N, Scott CR, Torra R, Tuffaha A, Jovanovic A, Waldek S, Packman S, Ludington E, Viereck C, Kirk J, Yu J, Benjamin ER, Johnson F, Lockhart DJ, Skuban N, Castelli J, Barth J, Barlow C, Schiffmann R. Treatment of Fabry's Disease with the Pharmacologic Chaperone Migalastat. N Engl J Med. 2016 Aug 11;375(6):545-55. doi: 10.1056/NEJMoa1510198. PMID 27509102
- [Background] Biegstraaten M, Arngrimsson R, Barbey F, Boks L, Cecchi F, Deegan PB, Feldt-Rasmussen U, Geberhiwot T, Germain DP, Hendriksz C, Hughes DA, Kantola I, Karabul N, Lavery C, Linthorst GE, Mehta A, van de Mheen E, Oliveira JP, Parini R, Ramaswami U, Rudnicki M, Serra A, Sommer C, Sunder-Plassmann G, Svarstad E, Sweeb A, Terryn W, Tylki-Szymanska A, Tondel C, Vujkovac B, Weidemann F, Wijburg FA, Woolfson P, Hollak CE. Recommendations for initiation and cessation of enzyme replacement therapy in patients with Fabry disease: the European Fabry Working Group consensus document. Orphanet J Rare Dis. 2015 Mar 27;10:36. doi: 10.1186/s13023-015-0253-6. PMID 25885911
- [Background] Ortiz A, Germain DP, Desnick RJ, Politei J, Mauer M, Burlina A, Eng C, Hopkin RJ, Laney D, Linhart A, Waldek S, Wallace E, Weidemann F, Wilcox WR. Fabry disease revisited: Management and treatment recommendations for adult patients. Mol Genet Metab. 2018 Apr;123(4):416-427. doi: 10.1016/j.ymgme.2018.02.014. Epub 2018 Feb 28. PMID 29530533
- [Background] Zarate YA, Hopkin RJ. Fabry's disease. Lancet. 2008 Oct 18;372(9647):1427-35. doi: 10.1016/S0140-6736(08)61589-5. PMID 18940466